CLINICAL TRIAL: NCT05403801
Title: Harnessing Mobile Technology to Deliver Tailored, Brief Pain-CBT for Advanced Cancer Patients on Opioids for Pain
Brief Title: STAMP+CBT mHealth for Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Palliative Care Research Center (Other)
Responsible Party: Principal Investigator, Desiree R. Azizoddin PsyD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-719
Record Dates: First submitted 2022-05-26; First posted 2022-06-03 (Actual); Results first posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-11

CONDITIONS: Active Cancer; Active Cancer Treatment; Advanced Cancer; Palliative Care; Chronic Pain Due to Cancer
Keywords: Active cancer; Active cancer treatment; Advanced Cancer; Palliative care; Chronic Pain due to Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STAMP+CBT PILOT (Experimental): Patients in this Pilot Cohort will be in the research study for 6 weeks total including:
  * a 4-week intervention period and 2-week post intervention period.
  * Patients will use the app for a total of 4 weeks (4-week intervention period), and will complete surveys at baseline, 4 weeks (end of intervention period), and at 6 weeks (end of 2-week post intervention period).
  Interventions: Behavioral: STAMP+CBT application

INTERVENTIONS:
Behavioral: STAMP+CBT application — Use the STAMP+CBT mobile app for 4 weeks (intervention period, 4 weeks for content introduction, extended 2 weeks for review of content if patient's request this

SUMMARY:
The purpose of this study is to test whether a mobile application developed to help people with cancer pain is useful and helpful to patients with cancer.

DETAILED DESCRIPTION:
This research study involves the use of a smartphone app at home in addition to surveys and potentially an interview at the end of the study.

The research study procedures include screening for eligibility, study interventions include surveys at the beginning of the study, after 4 weeks, and after 6 weeks and use of the smartphone app.

Participants will be on this research study for up to 6 weeks.

It is expected that about 15 people will take part in this research study

This research study is a Feasibility Study, which is the first-time investigators are examining this mobile application meant to help participant to learn behavioral techniques to manage cancer pain. The purpose is to make sure the app is usable and helpful for patients with cancer, and to get feedback about patient experiences after using the app for four weeks.

ELIGIBILITY:
Inclusion Criteria:

- PILOT COHORT

* Age ≥ 18 years
* Patients diagnosed with an active cancer diagnosis, either undergoing active cancer treatment or receiving treatment for an advanced cancer or are receiving palliative care
* Treatment managed at participating clinic (DFCI outpatient palliative care, gastrointestinal cancer center, and DFCI satellite clinic Merrimack Valley or Londonderry)
* Chronic pain related to cancer or treatment (> pain score of 4)
* Has an active prescription for at least one opioid medication to treat their cancer pain (i.e. not for post-surgical pain)
* Own a compatible smartphone (android) or is willing to use an android device provided by the study team
* Completes baseline survey

Exclusion Criteria:

* Patients in survivorship: patients who have completed their treatment regimens, are not actively receiving treatment for an advanced cancer, or have a cancer that is in remission
* Cognitive impairment that would interfere with study participation, as judged by treating clinician
* Inability to speak English: the intervention has not yet been translated to Spanish
* History of opioid use disorders
* Enrolled in hospice
* Currently hospitalized
* Use of transmucosal fentanyl, given safety concerns and ongoing risk mitigation program required to prescribe these (TIRF REMS).
* Pain primarily related to a recent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desiree Azizoddin, PsyD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber at Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber at Londonderry, Londonderry, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Azizoddin DR, DeForge SM, Baltazar A, Edwards RR, Allsop M, Tulsky JA, Businelle MS, Schreiber KL, Enzinger AC. Development and pre-pilot testing of STAMP + CBT: an mHealth app combining pain cognitive behavioral therapy and opioid support for patients with advanced cancer and pain. Support Care Cancer. 2024 Jan 22;32(2):123. doi: 10.1007/s00520-024-08307-7. PMID 38252172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from outpatient palliative care clinics
Groups:
- Pilot Cohort: Patients will use the STAMP+CBT app for 4 weeks (or 6 weeks if they request to review content further). During this 4 week intervention period participants will engage in pain CBT content including a goal-setting module, relaxation exercises, and reviewing educational content on cancer pain and psychological concepts. Patients will also use the app daily to report symptoms or pain, catastrophizing, mood, and sleep, and their usage of prescribed opioid medications. Patients will complete survey assessments at baseline, 4 weeks (end of intervention period), and 6 weeks (end of 2-week post intervention period) assessing feasibility, acceptability, and usability of the of the STAMP+CBT app.
Period: Overall Study
Arm/Group | Pilot Cohort
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pilot Cohort
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Intervention Adherence Rate
Description: >70% of subjects complete >4 of the 6 pain-CBT modules and patients will complete 50% of surveys by the end of 4 weeks (completion of the 4-week intervention study period)
Time Frame: 4 Weeks
Population: Participants who tested the app for 4 weeks (n=8) completed daily their daily EMA surveys.
Measure: Mean (Standard Deviation); unit: EMA App Surveys
Units Other Than Participants: Total EMA App Surveys
Arm/Group | Pilot Cohort
Number analyzed (Participants) | 8
Number analyzed (Total EMA App Surveys) | 28
EMA App Surveys | 15.75 (6.76)

2. Primary Outcome: Acceptability Rate
Description: Participants completed a modified version of the Acceptability E-scale, rating the app on a 5-point Likert scale (1-5), across 5 unique items on the following 5 domains: understandability, enjoyability, ease of use, time required to use it, and overall satisfaction.[Tariman, 2011] Higher scores indicated greater acceptability. Acceptability was pre-defined as >80% across all acceptability items rated as >4 or higher out of 5. Acceptability was evaluated by determining the mean score of all items for all participants (range of scale of score 1-5).
Time Frame: 4 weeks
Population: Evaluate each acceptability items that were rated as 4 or higher out of 5 for all patients
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pilot Cohort
Number analyzed (Participants) | 8
scores on a scale | 4.26 (1.07)

3. Secondary Outcome: Number of Enrolled Participants Who Consented and Completed the Study
Description: Participants were defined as individuals who consented and enrolled in the trial and completed 28 days of app use and completed study measures.
Time Frame: 7 Months
Population: 10 patients were recruited in 7 months and 8 remained in the study and completed all study activities and measures.
Measure: Number; unit: participants
Groups:
- Pilot Cohort: Patients will use the STAMP+CBT app for 4 weeks (or 6 weeks if they request to review content further). During this 4 week intervention period participants will engage in pain CBT content including a goal-setting module, relaxation exercises, and educational content. Patients will also use the app daily to report symptoms or pain, catastrophizing, mood, and sleep, and their usage and satisfaction of painkiller or prescribed medications. Patients will complete survey assessments at baseline, 4 weeks (end of intervention period), and 6 weeks (end of 2-week post intervention period) assessing pain severity, self-efficacy and catastrophizing, physical function, opioid use, and quality of life outcomes. Patients will lastly have an end-of-intervention interview assessing usability and acceptability of the STAMP+CBT app.
Arm/Group | Pilot Cohort
Number analyzed (Participants) | 10
participants | 8

4. Secondary Outcome: Study Retention
Description: The goal of the study was to have 60% of patients who enroll to the app will complete app use (use the app for 28 days) at the end of the 4 weeks and surveys at 4 and 6 weeks after enrollment
Time Frame: 6 Months
Population: Percent of patients who consented and also completed 4 weeks of app use and surveys at 4 and 6 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Cohort
Number analyzed (Participants) | 10
Participants | 8

5. Secondary Outcome: COMPREHENSIVE ENDPOINT
Description: Overall acceptability will be determined based on composite evaluation of acceptability ratings using the modified items from the Acceptability E-Scale [Tariman 2011]. Participants completed a modified version of the Acceptability e-scale, rating the app on a 5-point Likert scale on the following 5 domains: understandability, enjoyability, ease of use, time required to use it, and overall satisfaction. Higher scores indicated higher acceptability. Acceptability was pre-defined as >80% of all acceptability items being rated individually as >4 out of 5 (possible scores on this scale range between 1-5). Acceptability was evaluated by determining the mean score on each item individually, across all participants (range of scale of score 1-5).
Time Frame: 6 Weeks
Population: Patients rated the app's perceived acceptability on understandability, enjoyability, ease of use, time required to use it, and overall satisfaction on a 5-point Likert scale.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Pilot Cohort
Number analyzed (Participants) | 8
scores on a scale
  Ease of use | 4.29 (0.45)
  Understandability | 5.0 (0)
  Enjoyability | 4.14 (0.64)
  Time acceptability | 4.14 (0.99)
  overall Satisfaction | 4.29 (0.45)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Pilot Cohort
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT05403801/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT05403801/ICF_001.pdf